CLINICAL TRIAL: NCT01432834
Title: Evaluation of the Efficacy of the Allegretto Wave and the Wavefront Optimized Ablation Profile in Non-anterior Astigmatisms
Brief Title: Efficacy of the Wavefront Optimized (WFO) Profile in Non-anterior Astigmatisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Senior Lecturer of Ophthalmology, Democritus University of Thrace
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23/29-07-11
Record Dates: First submitted 2011-09-12; First posted 2011-09-13 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Astigmatism
Keywords: non-anterior astigmatism correction; Allegretto Wave excimer laser; wavefront optimized ablation profile (WFO); LASIK; PRK
MeSH Terms: conditions — Astigmatism | interventions — Keratomileusis, Laser In Situ; Photorefractive Keratectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LASIK group (LG group) (Other): Volunteers of this group received LASIK treatment.
  Interventions: Other: Laser in situ keratomileusis (LASIK)
- PRK group (PG group) (Other): Volunteers of this group received PRK treatment
  Interventions: Other: Photorefractive keratectomy (PRK)

INTERVENTIONS:
Other: Laser in situ keratomileusis (LASIK) — During LASIK treatments the Carriazo-Pendular microkeratome (SCHWIND eye-tech-solutions GmbH & Co.KG, Kleinostheim, Germany) with 130μm cutting head was used for the creation of the flap. The normal value of the negative pressure of the suction ring was between 600-620 mmHg and the velocity of the head movement was constant (3mm/sec). The hinge was created at the 12 o'clock position. The Allegretto Wave excimer laser (software version: 2.020 / WaveLight AG, Erlangen, Germany) was used for all ablations. Attempted ablations were modified according to the "S001 Wellington" nomogram for the "wavefront optimised" protocol.
  Other Names: Allegretto Wave excimer laser (software version: 2.020 / WaveLight AG, Erlangen, Germany); Carriazo-Pendular microkeratome (SCHWIND eye-tech-solutions GmbH & Co.KG, Kleinostheim, Germany)
  Arms: LASIK group (LG group)
Other: Photorefractive keratectomy (PRK) — The same surgical procedure was applied to all PG participants that included: Instillation of proparacaine hydrochloride 0.5% drops for topical anaesthesia, application of a sponge saturated with 10% alcohol to the central cornea for 20-30 seconds and subsequent de-epithelialization by means of a hockey knife.The Allegretto Wave excimer laser (software version: 2.020 / WaveLight AG, Erlangen, Germany) was used for all ablations. Attempted ablations were modified according to the "S001 Wellington" nomogram for the "wavefront optimised" protocol. A soft therapeutic lens was applied until complete re-epithelialization of the cornea was detected.
  Other Names: Allegretto Wave excimer laser (software version: 2.020 / WaveLight AG, Erlangen, Germany)
  Arms: PRK group (PG group)

SUMMARY:
The purpose of the study was to assess the efficacy of the Allegretto Wave excimer laser and the wavefront optimized ablation profile in correcting primarily non-anterior astigmatism faults, following laser in-situ keratomileusis (LASIK) and photorefractive keratectomy (PRK).

DETAILED DESCRIPTION:
Different optical components of the eye contribute to the total astigmatism error.In specific, the anterior corneal surface is responsible for the anterior component of astigmatism fault (anterior astigmatism), while the posterior corneal surface and the lens are responsible for the posterior one (posterior astigmatism).

Regarding our study, 74 refractive surgery candidates were recruited. Only one eye from each candidate was randomly enrolled in the study. Of them, 40 eyes underwent LASIK treatment (LG group), while 34 eyes underwent PRK treatment (PG group). The Allegretto Wave excimer laser (software version: 2.020 / WaveLight AG, Erlangen, Germany) was used for the ablation in all groups. Preoperatively, the ocular residual astigmatism (ORA) was calculated for each eye, according to which each astigmatism fault was characterized as primarily anterior or non-anterior.ORA is the vectorial value of astigmatism arising from non-anterior sources. Its amount on total astigmatism (R) is determined by the magnitude ratio ORA/R. Ratios below 1 indicate primarily anterior astigmatism, while ratios above 1 indicate primarily non-anterior astigmatism. 20 LG eyes and 16 PG eyes presented primarily anterior astigmatism (LG-A and PG-A subgroups, respectively), while 20 LG eyes and 18 PG eyes demonstrated primarily non-anterior astigmatism (LG-NA and PG-NA subgroups, respectively). Postoperatively, vector analysis of astigmatism correction was conducted; The following indexes were calculated: a) Correction index (CI), b) Difference vector (DV) and c) Index of Success (IOS).

ELIGIBILITY:
Inclusion Criteria:

* astigmatism fault

Exclusion Criteria:

* previous incisional eye surgery
* evidence of any type of corneal pathology
* evidence of any type of optic neuropathy
* history of optic neuropathy
* diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2010-04; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
vector analysis of astigmatism correction, following laser in-situ keratomileusis (LASIK) & photorefractive keratectomy (PRK) treatments. | 6 months postoperatively
  Vector analysis of astigmatism correction was conducted using preoperative and 6-month postoperative data. The following indexes were calculated: a) Correction index (CI) which is determined by the ratio of the surgically induced astigmatism (SIA) to the target induced astigmatism (TIA), b) Difference vector (DV) as an absolute measure of success, and, c) Index of Success (IOS) which is determined by the relationship of the DV to the TIA, as a relative measure of success.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Institute of Thrace (EIT), Alexandroupoli, Greece

REFERENCES:
- [Result] Labiris G, Gatzioufas Z, Giarmoukakis A, Sideroudi H, Kozobolis V. Evaluation of the efficacy of the Allegretto Wave and the Wavefront-optimized ablation profile in non-anterior astigmatisms. Acta Ophthalmol. 2012 Sep;90(6):e442-6. doi: 10.1111/j.1755-3768.2012.02463.x. Epub 2012 Jun 13. PMID 22690672